CLINICAL TRIAL: NCT03780816
Title: Variation in Cancer Centers' End-of-Life Quality
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Amber Barnato, Principal Investigator, Dartmouth-Hitchcock Medical Center
Other Study IDs: D18149
Record Dates: First submitted 2018-11-09; First posted 2018-12-19 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pilot Site: Norris Cotton Cancer Center: Observation and interview protocols will be piloted at this site. The content of these observations and interviews will not be analyzed for content.
  Interventions: Other: Observation of provider-patient interactions and interviews
- Karmanos Cancer Institute: Observations and interviews will be analyzed to identify any emergent concepts, categories, and relationships in the data.
  Interventions: Other: Observation of provider-patient interactions and interviews
- UNC Lineberger Comprehensive Cancer Center: Observations and interviews will be analyzed to identify any emergent concepts, categories, and relationships in the data.
  Interventions: Other: Observation of provider-patient interactions and interviews
- UAB O'Neal Comprehensive Cancer Center: Observations and interviews will be analyzed to identify any emergent concepts, categories, and relationships in the data.
  Interventions: Other: Observation of provider-patient interactions and interviews

INTERVENTIONS:
Other: Observation of provider-patient interactions and interviews — Clinical interactions between cancer patients and providers will be observed and hand-written field notes recorded and later transcribed. Semi-structured interviews with providers, patients, caregivers, and other informants will take place following initial observation.

SUMMARY:
This is a qualitative study of local organizational and provider practice norms, and how these norms influence patient and family expectations and provider decision-making heuristics for minority patients with advanced cancer at major US cancer centers. Outpatient visits with oncologists will be observed and documented via hand-written field notes. Semi-structured interviews with selected participating clinicians, patients, caregivers, and other informants will follow the initial observation.

DETAILED DESCRIPTION:
The purpose of this study is to identify organizational and provider practice norms at major US cancer centers, and how these norms influence patient and family expectations and provider decision-making heuristics for later-line chemotherapy, hospice, and ICU admission among minority patients with advanced cancer. Norms are rules about which there is at least some degree of consensus, enforced through social sanctions. Heuristics are unconscious judgments or rules of thumb.The study team will collect direct observation data from outpatient clinic visits, and semi-structured interview data from selected participating providers, patients, caregivers, and other informants following the initial observation.

The study team will perform 2-week, qualitative case studies of 3 theoretically sampled National Comprehensive Cancer Network (NCCN) and NCI Comprehensive Cancer Centers. Oncology practice managers' nominations of providers with particular cancer focuses, high volumes, and high peer influence will be used to sample oncologic clinicians to shadow in outpatient clinic settings. Observations will be hand-written during the clinic visit, and later dictated and transcribed. Observed providers will be invited to be interviewed. Select patients and caregivers will also be invited to be interviewed following initial clinic observation. Other informants will be invited to be interviewed on an ad hoc basis. All interviews will be audio recorded and transcribed, and interviews will be semi-structured to allow for natural flow of conversation. Observations and interviews will all be done by the study PI, project coordinator, and/or another research team member.

Clinical observations and semi-structured interviews will assess the following outcomes: 1) formal and informal organizational norms influencing provider decision-making, 2) provider decision-making heuristics, and 3) patient and caregiver expectations. All outcomes will be assessed regarding receipt of chemotherapy in the last 14 days of life, intensive care unit (ICU) admission in the last 30 days of life, and non or late hospice referral.

The investigators aim to to explore the how COVID-19 intersects with organizational and provider norms, practices, and service delivery for patients with advanced cancer.

ELIGIBILITY:
Provider Inclusion Criteria:

* Hospital-based providers (e.g., hospitalists, intensivists, emergency medicine, advanced practice providers) or oncology providers (e.g. medical oncologists, radiation oncologists, surgical oncologists, advanced practice providers)
* Care for patients with advanced cancer
* High clinical load
* Have high peer influence

Patient Inclusion Criteria:

* Advanced cancer
* Provider "would not be surprised" if patient died in the next 12 months

Caregiver Inclusion Criteria:

-Self-reported caregiver of a patient meeting inclusion criteria

Other Informant Inclusion Criteria:

- Member of the cancer center, hospital, unit, or service line leadership

Patient Exclusion Criteria:

- Potential medical malpractice cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatient and inpatient oncology providers who meet inclusion criteria and are nominated by their practice managers will be observed. If providers do not opt out after being introduced to the study by cancer center leadership, providers will be contacted directly for recruitment. A sub-sample of observed providers will be invited to participate in semi-structured interviews.
  A sub-sample of all patients (and caregivers) cared for by the shadowed provider who meet inclusion criteria will be invited to participate in semi-structured interviews. Recruitment will seek equal numbers of minority and non-minority participants.
  Personnel involved in developing and enforcing organizational policies, procedures, and practices, will also be invited to participate in semi-structured interviews.
Sampling Method: Non-Probability Sample
Enrollment: 473 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Formal and informal norms influencing provider decision making as assessed using ethnographic observation | 2-week site observation period
  Formal and informal norms influencing provider decision making (regarding receipt of chemotherapy in the last 14 days of life, intensive care unit (ICU) admission in the last 30 days of life, and non or late hospice referral) will be assessed using ethnographic observation in outpatient oncology clinics, multidisciplinary tumor boards, emergency departments, inpatient units, and other appropriate settings. All observations will be hand-written and later transcribed. Observations will be coded using an a priori framework, and subjected to thematic analysis.
Provider decision making heuristics as assessed using ethnographic observation | 2-week site observation period
  Provider decision making heuristics (regarding receipt of chemotherapy in the last 14 days of life, intensive care unit (ICU) admission in the last 30 days of life, and non or late hospice referral) will be assessed using ethnographic observation in outpatient oncology clinics, multidisciplinary tumor boards, emergency departments, inpatient units, and other appropriate settings. All observations will be hand-written and later transcribed. Observations will be coded using an a priori framework, and subjected to thematic analysis.
Patient expectations as assessed using ethnographic observation | 2-week site observation period
  Patient expectations (regarding receipt of chemotherapy in the last 14 days of life, intensive care unit (ICU) admission in the last 30 days of life, and non or late hospice referral) will be assessed using ethnographic observation in outpatient oncology clinics, emergency departments, inpatient units, and other appropriate settings. All observations will be hand-written and later transcribed. Observations will be coded using an a priori framework, and subjected to thematic analysis.
Formal and informal norms influencing provider decision making as assessed using semi-structured interviews | 2-week site observation period
  Formal and informal norms influencing provider decision making (regarding receipt of chemotherapy in the last 14 days of life, intensive care unit (ICU) admission in the last 30 days of life, and non or late hospice referral) will be assessed using a study-specific semi-structured interview, with all interviews audio recorded and transcribed, coded using an a priori framework, and subjected to thematic analysis.
Provider decision making heuristics as assessed using semi-structured interviews | 2-week site observation period
  Provider decision making heuristics (regarding receipt of chemotherapy in the last 14 days of life, intensive care unit (ICU) admission in the last 30 days of life, and non or late hospice referral) will be assessed using a study-specific semi-structured interview, with all interviews audio recorded and transcribed, coded using an a priori framework, and subjected to thematic analysis.
Patient expectations as assessed using semi-structured interviews | 2-week site observation period
  Patient expectations (regarding receipt of chemotherapy in the last 14 days of life, intensive care unit (ICU) admission in the last 30 days of life, and non or late hospice referral) will be assessed using a study-specific semi-structured interview, with all interviews audio recorded and transcribed, coded using an a priori framework, and subjected to thematic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Amber E Barnato, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knutzen KE, Schifferdecker KE, Murray GF, Alam SS, Brooks GA, Kapadia NS, Butcher R, Barnato AE. Role of norms in variation in cancer centers' end-of-life quality: qualitative case study protocol. BMC Palliat Care. 2020 Aug 27;19(1):136. doi: 10.1186/s12904-020-00641-x. PMID 32854691